CLINICAL TRIAL: NCT05494086
Title: Dual-Port Laparoscopic Distal Gastrectomy for Gastric Cancer: A Randomised Clinical Trial
Brief Title: Dual-Port Laparoscopic Distal Gastrectomy for Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-266
Record Dates: First submitted 2022-07-10; First posted 2022-08-09 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: DPLDG group :Reduced Port Laparoscopic Distal Gastrectomy LDG group: Laparoscopic Distal Gastrectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPLDG arm (Experimental): Dual-port laparoscopic distal gastrectomy
  Interventions: Procedure: DPLDG
- LDG arm (Active Comparator): Laparoscopic distal gastrectomy
  Interventions: Procedure: LDG

INTERVENTIONS:
Procedure: DPLDG — Dual-port laparoscopic distal gastrectomy
  Arms: DPLDG arm
Procedure: LDG — Laparoscopic distal gastrectomy
  Arms: LDG arm

SUMMARY:
Dual-port laparoscopic gastrectomy (DPLG) has been widely performed in recent years for treating gastric cancers. The present study explore the safety and effect of dual-port laparoscopic distal gastrectomy (DPLDG).

DETAILED DESCRIPTION:
As a novel minimally invasive technique,laparoscopic surgery has presently become widely accepted as an alternative treatment for malignant diseases. In the treatment of gastric cancers, it has been reported to be an optionalprocedure with the advantages of less invasiveness,less blood loss, faster postoperative recovery and shorter hospital stay, when compared to open surgery. In general, four or five trocars are required in conventional laparoscopic distal gastrectomy (CLDG), and each port results in abdominal injury, which may lead to port site complications, such as wound infection, dehiscence and small bowel herniation. Hence, it remains challenging to determine whether surgical wounds could be minimized during laparoscopic gastric surgery. The development of reduced-port laparoscopic techniques has been largely due to the appearance of multi-channel ports. A conventional trocar port can only be used for inserting a single instrument. With the advancement of laparoscopic devices, a variety of multi-channel ports have been introduced and used in laparoscopic surgeries. At present, multi-channel ports that have been reported include Uni-X devices (Pnavel Systems, Brooklyn, NY, USA), TriPort devices (Advanced Surgical Concepts,Wicklow, Ireland), SILS devices (Covidien, Norwalk, CT, USA), OctoPort devices (DalimSurgNet, Seoul, Korea) and self-made multichannel devices from medical centers globally. The number of ports located on these multichannel devices varies from two to four. Twoport and three-port devices are more commonly used at present in laparoscopic gastric cancer surgery. In recent years, the use of reduced-port laparoscopic gastrectomy has rapidly increased. Several studies have suggested that, in contrast to conventional laparoscopic gastrectomy (CLG), the reduced-port method has some apparent postoperative benefits in the treatment of gastric cancers, such as shorter hospital stay, less pain, less blood loss and better cosmetic results. Among these studies, most have been about distal gastrectomy. Hence, the application of this technique in total gastrectomy is at present relatively less. As a type of reduced-port technique, Kawamura et al. first used this technique in 2011 to treat early distal gastric cancers, and suggested that dual-port laparoscopic distal gastrectomy (DPLDG) is superior to conventional approaches from the cosmetic standpoint, and has the potential to become a technically acceptable procedure. However, due to the more limited operating space when compared to CLDG, it has been generally considered that DPLDG is more difficult to perform than CLDG. The difficulty of DPLDG is mainly due to insufficient intraoperative traction and exposure, which makes the principle of triangulation and counteraction in DPLDG less good when compared to those in CLDG. In addition, since merely one additional trocar is located at one side of the abdominal wall, it is difficult for the surgeon to change position with the assistant, when necessary. The application of DPLDG to distal gastric cancer remains controversial, and critical comments have been made regarding it.

ELIGIBILITY:
Inclusion Criteria:

1. patients within 18--75 years old;
2. patients with a preoperative pathological diagnosis of gastric adenocarcinoma;
3. patients with a clinical tumor stage of T1N1,T2N0 according to the preoperative examinations (gastroscopy, ultrasound gastroscopy and computed tomography);
4. patients with a plan to undergo laparoscopic distal gastrectomy and obtain R0 surgical results;
5. patients without severe heart, liver, lung, or kidney dysfunction;
6. patients with an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1; and (7) patients with American Society of Anesthesiologists (ASA) I-II.

Exclusion Criteria:

1. patients with a history of upperabdominal surgery;
2. patients who presentedas an emergency case;
3. patients with other histories of malignant diseases within 5 years;
4. patients with prior neoadjuvant chemotherapy or radiation therapy; and (5)patients who need simultaneous surgical treatment for other malignant diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Early operative morbidity | Within 30 days following surgery
  Including wound complications (infection, effusion, dehiscence,poor healing), intra-abdominal active bleeding,digestive tract active bleeding, anastomotic leakage, anastomotic stenosis, intestinal fistula, pancreatic fistula, chylous fistula, intra-abdominal abscess formation, gastroparesis, intestinal paralysis, intestinal obstruction, cholecystitis, pancreatitis, pneumonia, pleural effusion, pulmonary embolism, cardiocerebrovascular complications, deep venous thrombosis, urinary tract complications, catheter-related complications, condition of pain,etc.;

SECONDARY OUTCOMES:
5 year overall survival rate | 5 years
  From date of randomization until the date of first documented date of death from any cause, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University; Tian Lin, Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All
Supporting Information: Study Protocol, SAP
Access Criteria: All